CLINICAL TRIAL: NCT06907758
Title: Impact of Perioperative Organ Resuscitation of Brain-dead Deceased Organ Donor on Kidney Graft Function in the Recipient
Acronym: OPTI-PMO 2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9245
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Kidney Graft
Keywords: Kidney Graft; Grafts; Organ transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain-dead patients are the primary source of grafts for those awaiting organ transplantation. Recommendations exist for the management of these potential donors, based on the concept of organ resuscitation, according to which targeted resuscitation would improve graft quality and quantity.

Graft performance thus depends on fixed factors (donor/recipient age, medical history, etc.) but also potentially modifiable factors.

Through this study, the investigators aim to identify potentially modifiable factors in our donor care (in intensive care and the operating room) that may influence graft function in the recipient. For simplicity, the investigators will focus on kidney grafts. The aim is to improve the effectiveness of the transplant and reduce waiting times.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for organ donor patients are as follows:

* Adult patient
* Brain dead
* Hospitalized in surgical intensive care at Strasbourg University Hospital (NHC cardiovascular intensive care unit, NHC multi-purpose intensive care unit, Hautepierre surgical intensive care unit) from January 1, 2018 to December 31, 2023
* Having undergone multi-organ transplantation
* At least one of the donor kidneys has been transplanted to a patient at Strasbourg University Hospital
* Absence of written objection in the medical file of the subject (and/or their legal representative, if applicable) to the reuse of their data for scientific research purposes.

The inclusion criteria for kidney transplant recipients are as follows:

* Adult patient
* Recipient of a kidney transplant from an organ donor who meets the inclusion criteria for donor patients mentioned above
* Patient who has undergone surgery and is hospitalized post-operatively at Strasbourg University Hospital
* Patient monitored by the Strasbourg University Hospital transplant team
* Absence of written objection in the subject's medical file (and/or their legal representative, if applicable) to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject (and/or their legal representative, if applicable) who has expressed their opposition to the reuse of their data for scientific research purposes
* Brain-dead patient who has not undergone organ retrieval
* Brain-dead patient whose kidney has not been allocated to a recipient in Strasbourg
* Patient transferred to the Strasbourg University Hospital's intensive care unit from another hospital in a state of already diagnosed brain death solely for organ retrieval
* Kidney transplant patient with a graft from a living donor
* Kidney transplant patient with a graft from a deceased donor who is not brain-dead
* Kidney transplant patient with a graft from a deceased donor who is brain-dead and hospitalized in a hospital other than Strasbourg

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subject adulte
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Ratio of creatinine decrease | Days 1 and 2 in kidney transplant recipients
  Ratio of creatinine decrease on days 1 and 2 in kidney transplant recipients (formula: CRR2% = ((Cr1-Cr2)*100)/Cr1) or the need for dialysis before day 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie, Réanimation et Médecine Périopératoire - CHU de Strasbourg - France, Strasbourg, France